CLINICAL TRIAL: NCT03319446
Title: Collection of Anonymized Samples for Use in Product Development and Clinical Trials
Brief Title: Collection of Anonymized Samples
Status: Enrolling by invitation | Type: Observational
Sponsor: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DX-SDY-036556
Record Dates: First submitted 2017-10-18; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Healthy; Respiratory Disease; Gastrointestinal Disease
MeSH Terms: conditions — Respiration Disorders; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, rectal swabs, nasal washes, nasopharyngeal aspirates, nasopharyngeal swabs, throat swabs, nasal swabs, and urine from human sources.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a generic sample collection study for collecting blood, stool, rectal swabs, nasal washes, nasopharyngeal aspirates, nasopharyngeal swabs, throat swabs, nasal swabs, and urine from human sources. Subjects will be recruited from BioFire Diagnostics employees and from the general community. Subjects may be asked about recent or ongoing illness at the time of specimen collection and these symptoms will be recorded and attached to the sample. No other identifying information will be collected and the samples will be kept anonymous.The samples may be used internally or by external sites, such as the clinical study sites, for evaluating and determining performance characteristics of in vitro diagnostic devices.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult

Exclusion Criteria:

* Weigh less that 110 lb for blood collection

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Employees of BioFire Diagnostics, and the general community of the greater Salt Lake City area.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
PCR Amplification Curves | 10 years
  PCR amplification curves will be used to confirm the presence or absence of target analytes.

CONTACTS AND LOCATIONS:
Locations (1):
- BioFire Diagnostics, Salt Lake City, Utah, United States